CLINICAL TRIAL: NCT03632200
Title: Improvement of the Nutritional Course of Care After Surgical Treatment at the Patients Affected by a Cancer of the Head and by the Neck
Brief Title: Nutritional Course of Care After Surgical Treatment at the Patients Affected by a Cancer of the Head and by the Neck
Acronym: NUTRIMAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2018_843_0015
Record Dates: First submitted 2018-07-16; First posted 2018-08-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Nutrition Disorders; Head and Neck Cancer
MeSH Terms: conditions — Nutrition Disorders; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: a pilot study to compare experimental group (improved coverage) and control group (classic coverage)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patients with a cancer of the VADS: in preoperative, all the patients will benefit from dietary advice during a multidisciplinary specific consultation (physiotherapist, dietician, nursing staff CMF). The accent will be put on the adaptations of the diet, the complementary nutritional contributions, the assistants in "better to eat".
  In post-operative, a dietetic consultation will be set up in 7 days at the post hospitalization and rate call phone at M1, M2, M4 and M5.
  The undernourished patient will benefit besides a multidisciplinary consultation at the rate of a consultation a month during 6 months according to the same conditions.
  Interventions: Other: Experimental group
- Control group (No Intervention): The patients will be followed according to the current recommendations of the French Society Clinical Nutrition and Metabolism (SFNEP).

INTERVENTIONS:
Other: Experimental group — The patients with a cancer of the VADS: in preoperative, all the patients will benefit from dietary advice during a multidisciplinary specific consultation (physiotherapist, dietician, nursing staff CMF). The accent will be put on the adaptations of the diet, the complementary nutritional contributions, the assistants in "better to eat".
  In post-operative, a dietetic consultation will be set up in 7 days at the post hospitalization and rate call phone at M1, M2, M4 and M5.
  The undernourished patient will benefit besides a multidisciplinary consultation at the rate of a consultation a month during 6 months according to the same conditions
  Other Names: multidisciplinary specific consultation
  Arms: Experimental group

SUMMARY:
Whatever are the strategies of coverage, the consideration of the state of bad nutrition is not often the priority. According to the last recommendations (2012) of the French Society Clinical Nutrition and Metabolism (SFNEP), the surgeries of the cancers of the VADS are not listed among surgeries with high morbidity. So the specific recommendations for the patients undernourished with surgery with low morbidity, only a personalized dietary advice and oral nutritional supplements are recommended in preoperative. There is no specific recommendation in post-operative.

Two groups of cancer patients of the VADS will be compared: a control group benefiting from a nutritional coverage based on the current recommendations of the SFNEP, an experimental group benefiting from an improved nutritional coverage.

In preoperative, all the patients of experimental group will benefit from dietary advice during a multidisciplinary specific consultation. In post-operative, a dietetic consultation will be set up in 7 days at the exit of hospitalization and call phone at M1, M2, M4 and M5. And for the undernourished patient will benefit a multidisciplinary consultation at the rate of a consultation a month during 6 months.

In the Group control, the patients will be followed according to the current recommendations of the SFNEP.

DETAILED DESCRIPTION:
Whatever are the strategies of coverage, the consideration of the state of bad nutrition is not often the priority. According to the last recommendations (2012) of the French Society Clinical Nutrition and Metabolism (SFNEP), the surgeries of the cancers of the VADS are not listed among surgeries with high morbidity. So the specific recommendations for the patients undernourished with surgery with low morbidity, only a personalized dietary advice and oral nutritional supplements are recommended in preoperative. There is no specific recommendation in post-operative.

Two groups of cancer patients of the VADS will be compared: a control group benefiting from a nutritional coverage based on the current recommendations of the SFNEP, an experimental group benefiting from an improved nutritional coverage.

In preoperative, all the patients of experimental group will benefit from dietary advice during a multidisciplinary specific consultation. In post-operative, a dietetic consultation will be set up in 7 days at the exit of hospitalization and call phone at M1, M2, M4 and M5. And for the undernourished patient will benefit a multidisciplinary consultation at the rate of a consultation a month during 6 months.

In the Group control, the patients will be followed according to the current recommendations of the SFNEP.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by a cancer of the VADS
* Man or woman of 18 and more years old
* Patient benefiting from a surgery for its cancer of the VADS
* Patient having signed a written consent
* Patient member in a national insurance scheme

Exclusion Criteria:

* Patient minor
* Patient benefiting from a radiotherapy
* Patient participant in another research interfering on the nutritional state of the patient
* Patients under guardianship or guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The satisfactory nutritional state defined by the absence of loss of weight | 6 months
  weight loss difference equal to 0 between the time 0 and the 6th month

SECONDARY OUTCOMES:
The score PG-SGA (index of Detsky) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Dakpé, MD, Principal Investigator — CHU Amiens Picardie
Locations (1):
- CHU Amiens-Picardie, Amiens, France